CLINICAL TRIAL: NCT01993901
Title: The Influence of Clinical Specialist Radiation Therapist (CSRT)-Led Telephone Follow-up on Edmonton Symptom Assessment Scale (ESAS) Scores in Patients Who Have Been Treated With Lung Stereotactic Body Radiation Therapy (SBRT)
Brief Title: The Influence of CSRT-led Telephone Follow-up on ESAS Scores in Patients Who Have Been Treated With Lung SBRT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never officially opened
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Darby Erler, Clinical Specialist Radiation Therapist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PBR041575
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Lung Cancer, Anxiety Post SBRT
Keywords: lung SBRT, ESAS, anxiety
MeSH Terms: conditions — Lung Neoplasms; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSRT led telephone follow up (Experimental): Patients in the experimental arm will be telephoned by the CSRT 4-6 weeks after completion of their treatment to assess any symptoms.
  Interventions: Other: CSRT led telephone follow up
- Standard Follow up (No Intervention): Patients in the control group will have the standard follow up (CT of the chest, abdomen and pelvis prior to follow-up with the radiation oncologist 4 months after the completion of their treatment). In order to control for an "attention effect" that may be seen in the intervention group, patients in the control group will get a placebo or sham telephone call initiated by a research assistant 4-6 weeks after completion of their treatment. This telephone call will simply confirm their follow up appointment.

INTERVENTIONS:
Other: CSRT led telephone follow up — Patients in the intervention group will be telephoned by the CSRT 4-6 weeks after completion of their treatment to assess any symptoms. A second follow up telephone call will be made at 12 weeks post treatment if required in order to address treatment related side effects that were identified during the first call and any interventions that were recommended
  Arms: CSRT led telephone follow up

SUMMARY:
The principal aim of this study is to prospectively assess if Clinical Specialist Radiation Therapist (CSRT) led telephone follow up after treatment with lung Stereotactic Body Radiation Therapy (SBRT) has an impact on patient symptom burden as assessed by Edmonton Symptom Assessment Scale (ESAS) scores.

DETAILED DESCRIPTION:
Design:

The design of this study is a randomized control trial. The study population will include patients treated with lung SBRT at Sunnybrook Odette Cancer Centre (OCC) over a specified 1 year time period who have consented to participating in the study.

Methods:

Patients who consent to the study will be randomized into either the control group or intervention group. Simple randomization will be completed using a computer-generated random number table. Baseline ESAS scores will be collected on the last day of radiation treatment for both groups. Patients in the intervention group will be telephoned by the CSRT 4-6 weeks after completion of their treatment to assess any symptoms. The CSRT will advise the patient on how to manage their side effects and address any anxieties the patient may feel based on published response care paths such as Cancer Care Ontario's Symptom Management Guide. Referrals to the attending radiation oncologist will be made if the patients response in the physical items of ESAS such as pain, nausea and shortness of breath increases to above 2 from their baseline or if they require medical management for a side effect such as esophagitis. If there is an increase in the emotional symptom scores to greater than 2, the CSRT will discuss supportive options and facilitate a referral to social work with the patients' permission. Each telephone call will be logged on a standard template. A second follow up telephone call will be made at 12 weeks post treatment if required in order to address treatment related side effects that were identified during the first call and any interventions that were recommended. When the patient returns to clinic for their first regularly scheduled follow-up appointment, ESAS will be completed as well as a questionnaire to assess their opinions regarding their follow up.

Patients in the control group will have the standard follow up plan as outlined earlier (CT of the chest, abdomen and pelvis prior to follow-up with the radiation oncologist 4 months after the completion of their treatment) and will be asked to complete a questionnaire to assess their opinions regarding follow up during their clinic appointment. In order to control for an "attention effect" that may be seen in the intervention group, patients in the control group will get a placebo or sham telephone call initiated by a research assistant 4-6 weeks after completion of their treatment. This telephone call will simply confirm their follow up appointment and should the patient bring up any issues, they will be referred to the appropriate nursing telephone line.

Inclusion criteria:

• Any patient treated with lung SBRT over a specified one year time frame.

Exclusion criteria:

1. Patients who are not 18 years of age or greater
2. Patients whose first language is not English and require translation.
3. Patients who have poor hearing and find it difficult to carry on a telephone conversation.

ELIGIBILITY:
Inclusion Criteria:

* Any patient treated with lung SBRT over a specified one year time frame

Exclusion Criteria:

* Patients who are not 18 years of age or greater
* Patients whose first language is not English and require translation.
* Patients who have poor hearing and find it difficult to carry on a telephone conversation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Change in ESAS scores | 4 months after completion of SBRT
  Measure changes in ESAS scores in patients who have been treated with lung SBRT from the last day of treatment to the first follow up appointment

SECONDARY OUTCOMES:
Efficacy of CSRT led follow up | 4 months after completion of SBRT
  Determine if CSRT-led telephone led follow-up has an impact on the ESAS scores of patients treated with lung SBRT

OTHER OUTCOMES:
Patient opinions regarding follow up care | 4 months after SBRT
  Evaluate patients opinions regarding their follow up care

CONTACTS AND LOCATIONS:
Overall Officials: Lisa DiProspero, BSc, MSc, Study Director — Toronto Sunnybrook Regional Cancer Centre
Locations (1):
- Sunnybrook Odette Cancer Centre, Toronto, Ontario, Canada